CLINICAL TRIAL: NCT06736522
Title: Can A Youth Leadership and Mindfulness Program Support Well-being for Youth of Color?
Brief Title: Future Leaders Program: Testing a Youth Leadership, Engagement, and Mindfulness Program
Acronym: FLP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 7018E; 4UH3AT012530 (NIH)
Record Dates: First submitted 2024-12-12; First posted 2024-12-16 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Adolescent Behavior Problem; Mental Health Wellness 1
Keywords: mindfulness; youth leadership; youth wellbeing
MeSH Terms: interventions — Leadership; Mindfulness

STUDY DESIGN:
Intervention Model Description: Individually Randomized Group Treatment Trial Design
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be masked to study condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Leadership, Engagement, and youth Action Program with Mindfulness (Experimental): The Leadership, Engagement, and youth Action Program with Mindfulness intervention (LEAP) consists of 14 sessions focused on youth leadership and mindfulness.
  Interventions: Behavioral: Leadership, Engagement, and youth Action Program with Mindfulness
- EnvisionIT (Active Comparator): EnvisionIT is a college and career-readiness program designed for students in grades 6-12. The EnvisionIT program will be delivered over 14 sessions, and focus on skills and career/college readiness.
  Interventions: Behavioral: EnvisionIT

INTERVENTIONS:
Behavioral: Leadership, Engagement, and youth Action Program with Mindfulness — The Leadership, Engagement, and youth Action Program with Mindfulness intervention (LEAP) was designed and co-created with youth to improve youth well-being by enhancing leadership opportunities and by developing mindfulness in day-to-day life. LEAP seeks to foster these improvements in youth and to increase youth mental, emotional, and behavioral health. Youth voice is incorporated into the intervention, with facilitators leading the first 7 sessions, and youth leading the remainder.
  Other Names: LEAP
  Arms: Leadership, Engagement, and youth Action Program with Mindfulness
Behavioral: EnvisionIT — Participants in this arm will receive 14 sessions of EnvisionIT training, focused on preparing students with essential skills including digital literacy through competency in information technology, financial literacy, English language arts skills, and college and career readiness. All sessions will be delivered by facilitators trained in EnvisionIT.
  Arms: EnvisionIT

SUMMARY:
The current study tests the feasibility and effectiveness of a youth intervention designed to provide meaningful leadership opportunities through the acquisition of leadership skills as well as mindfulness practice, LEAP: Leadership, Engagement, and youth Action Program with Mindfulness.

The goal of this project is to determine whether the Leadership, Engagement, and youth Action Program with Mindfulness (LEAP) curriculum, which was developed with youth, is a feasible and effective intervention for fostering leadership and well-being. The investigators seek to understand whether LEAP can support wellbeing for youth as a strategy to increase youth mental, emotional, and behavioral (MEB) health.

DETAILED DESCRIPTION:
The LEAP study will determine whether a 14-session program designed to provide leadership and mindfulness skills to youth is an effective and feasible intervention. The curriculum consists of 14 two-hour sessions delivered after school. The comparison group will take part in EnvisionIT, a college and career readiness program designed for students in grades 6 through 12. EnvisionIT aims to prepare students with essential skills including digital literacy, and college and career readiness. The comparison group will also have 14 two-hour group sessions. Both LEAP and EnvisionIT will be delivered by trained facilitators. All participants in LEAP and EnvisionIT will be assessed at four time points; facilitators will also complete interviews post-intervention and provide feedback on data fidelity and acceptability following each session. This record reports on the UH3 phase of the grant.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents ages 14 and older in grades 9-12 during the Fall/Winter or in grades 9-11 during the Spring
* Enrolled in a partner site in Massachusetts or Illinois
* Adolescents are only included with parent consent and youth assent if they are under the age of 18. Adolescents at least 18 years old can provide consent.

Exclusion Criteria:

* They participated in the pilot phase (UG3)
* They cannot commit to participation in the full study (e.g., attendance at all intervention sessions)
* They are not in grades 9-12 at a partner site
* Parent/guardian has a preferred consent language other than English or Spanish.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 504 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Engagement, Perseverance, Optimism, Connectedness, and Happiness (EPOCH; Kern et al., 2016) measure of adolescent wellbeing | Baseline, 2-3 months, 6 months, 9 months
  20-item, 5-point scale measuring five positive characteristics that support higher levels of wellbeing: Engagement, Perseverance, Optimism, Connectedness, and Happiness. The scale range is 1-5, higher scores indicate better wellbeing.
Strengths and Difficulties Questionnaire (SDQ; Goodman, 2001) | Baseline, 2-3 months, 6 months, 9 months
  25 item multiple choice questionnaire that measures internalizing and externalizing problems and prosocial behavior (emotional, conduct, hyperactivity-inattention, peer, prosocial). The scale range is 0-40, higher scores indicate worse difficulties.
Self-Rated Health 12-item Short-Form Survey (SF-12; Ware et al., 1996) | Baseline, 2-3 months, 6 months, 9 months
  12 item 5-point survey measuring general health, asking about overall health self-rating, ability to do daily activities, energy levels, and physical and emotional limitations. The scale range is 0-100, higher scores indicate better health.

SECONDARY OUTCOMES:
Student Career Construction Inventory (Savickas, 2018) | Baseline, 2-3 months, 6 months, 9 months
  18 item measure 5-point survey measuring crystallizing a vocational self-concept, exploring to gather information about occupations, deciding to commit to an occupational choice, and preparing to implement that choice. Scale scores range from 1-5, with higher scores indicating greater focus on each of the four tasks of career choice construction.
Vocational Skills Self-Efficacy (VSSE; McWhirter et al., 2000) | Baseline, 2-3 months, 6 months, 9 months
  29 item 5-point survey measuring level of confidence to establish and work toward job goals. Scale scores range from 29-145, with higher scores indicating greater vocational self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Cruz-Gonzalez, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - University of Illinois, Chicago, Chicago, Illinois
  - METCO, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Determinations will be made on a case-by-case basis of what type of data can be shared while maintaining confidentiality of respondents. The investigators are still establishing a plan for data sharing.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be shared after findings for primary outcomes are published. Time frame for sharing will be based on requests, based on recommendations from the funding agency.
Access Criteria: Determinations will be made on a case-by-case basis of what type of data can be shared while maintaining confidentiality of respondents. Any data shared will be de-identified and will follow established systems for security in data use.

REFERENCES:
- [Background] Alegria M, Alvarez K, NeMoyer A, Zhen-Duan J, Marsico C, O'Malley IS, Mukthineni R, Porteny T, Herrera CN, Najarro Cermeno J, Kingston K, Sisay E, Trickett E. Development of a Youth Civic Engagement Program: Process and Pilot Testing with a Youth-Partnered Research Team. Am J Community Psychol. 2022 Mar;69(1-2):86-99. doi: 10.1002/ajcp.12548. Epub 2021 Aug 4. PMID 34350588